CLINICAL TRIAL: NCT02742493
Title: A Single-center, 3-arm, Parallel-group Randomized Controlled Trial to Evaluate the Effectiveness of Three Orthodontic Retention Schemes in Preventing Post-treatment Mandibular Arch Changes and Gingival Recession in Children and Adolescents
Brief Title: RCT for the Effectiveness of 3 Orthodontic Retention Schemes on Post-treatment Stability and Gingival Recession
Acronym: OrthRe10tion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Iosif Sifakakis, Associate Prof., Department of Orthodontics, School of Dentistry, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 294
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2025-01-14 (Actual); Status verified 2023-08

CONDITIONS: Relapse; Gingival Recession
Keywords: relapse; irregularity; recession; retention
MeSH Terms: conditions — Recurrence; Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0.028 bonded to canines (Experimental): lower fixed canine and canine retainer and upper removable Hawley (Intervention A)
  Interventions: Other: 0.028 bonded to canines
- 0.027 7-strand bonded to all 6 (Experimental): lower fixed canine to canine retainer and upper removable Hawley (Intervention B)
  Interventions: Other: 0.027 7-strand bonded to all 6
- removable Hawley-type (Active Comparator): lower hawley-type and upper hawley removable retainer (Control)
  Interventions: Other: removable Hawley-type

INTERVENTIONS:
Other: 0.028 bonded to canines — lower fixed canine and canine retainer (0.028 stainless steel bonded to canines) and upper removable Hawley (Intervention A)
  Arms: 0.028 bonded to canines
Other: 0.027 7-strand bonded to all 6 — lower fixed canine to canine retainer (7-strand Twistflex 0.027 bonded to all six anterior teeth) and upper removable Hawley (Intervention B)
  Arms: 0.027 7-strand bonded to all 6
Other: removable Hawley-type — lower Hawley-type and upper Hawley removable retainer (Control)
  Arms: removable Hawley-type

SUMMARY:
The present study aims to assess the effectiveness of three different retention schemes used to maintain tooth position after orthodontic treatment with fixed orthodontic appliances (stability) and to evaluate possible association between retention scheme and gingival recessions on the lingual surfaces of the lower anterior teeth seen for up to 5 years post-treatment. Moreover the possible association between primary relapse tendency and long term occlusal stability will be evaluated.

DETAILED DESCRIPTION:
This is a randomized, controlled, single-center, equivalence trial with three parallel groups and an allocation ratio of 1:1:1, that aims to investigate the effectiveness of 3 orthodontic retention schemes on post-treatment mandibular arch stability and gingival recession.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* Age between 10 and 16 years
* At the finishing stage of orthodontic treatment, programmed for debonding
* Class I to Class II molar relationship before the beginning of orthodontic treatment
* Non-extraction treatment plan with fixed straight-wire appliances
* Space deficiencies and irregularity of no more than 6mm in the maxillary/ mandibular arch (Irregularity Index)

Exclusion Criteria:

* No missing teeth, impacted teeth or other dental anomalies
* No congenital anomalies/ syndromes

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-03-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Little's Irregularity Index in the mandible (mm) | 1 year in retention, 2 years in retention, 5 years in retention
Changes in Intercanine width in the mandible (mm) | 1 year in retention, 2 years in retention, 5 years in retention
Changes in Interpremolar width in the mandible (mm) | 1 year in retention, 2 years in retention, 5 years in retention
Changes in Intermolar width in the mandible (mm) | 1 year in retention, 2 years in retention, 5 years in retention
Changes in Arch length in the mandible (mm) | 1 year in retention, 2 years in retention, 5 years in retention

SECONDARY OUTCOMES:
Changes in Gingival Recessions on the lingual surfaces of the six lower anterior teeth | 1 year in retention, 2 years in retention, 5 years in retention
Changes in Intercanine width in the maxilla (mm) | 1 year in retention, 2 years in retention, 5 years in retention
Changes in Interpremolar width in the maxilla (mm) | 1 year in retention, 2 years in retention, 5 years in retention
Changes in Intermolar width in the maxilla (mm) | 1 year in retention, 2 years in retention, 5 years in retention
Changes in Arch length in the maxilla (mm) | 1 year in retention, 2 years in retention, 5 years in retention
Changes in Overbite and Overjet (mm) | 1 year in retention, 2 years in retention, 5 years in retention
Accidental bond failures of fixed retainers or breakages of removable ones | 1 year in retention, 2 years in retention, 5 years in retention
Leveling or torque related problems of the lower anterior teeth | 1 year in retention, 2 years in retention, 5 years in retention

CONTACTS AND LOCATIONS:
Overall Officials: Iosif Sifakakis, Lecturer, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Department of Orthodontics, School of Dentistry, University of Athens, Athens, Goudi, Greece

IPD SHARING:
Plan to Share IPD: Yes